CLINICAL TRIAL: NCT04219579
Title: Continuous Versus Intermittent Infusion of Human Antithrombin III Concentrate in the Immediate Postoperative Period After Liver Transplantation
Brief Title: Antithrombin III Concentrate After Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Geol Ryu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HGRyu_AT-III
Record Dates: First submitted 2019-12-29; First posted 2020-01-07 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Liver Transplant; Complications
Keywords: antithrombin III; liver transplantation; administration method; dosage
MeSH Terms: interventions — Antithrombin III

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous infusion (Experimental): Immediately after operation, 2000 international unit (IU) of Antithrombin-III (AT-III) concentrate is loaded for 1 hour. AT-III concentrate 3000 IU is continuously infused through following 71 hours.
  Interventions: Drug: Antithrombin III, continuous infusion
- Intermittent infusion (Active Comparator): Every 6 hours, 500 IU of AT-III concentrate is infused through 1 hour during the first 72 hours after liver transplantation.
  Interventions: Drug: Antithrombin III, Intermittent infusion

INTERVENTIONS:
Drug: Antithrombin III, continuous infusion — Antithrombin-III is administered continuously
  Other Names: Antithrombin III, human
  Arms: Continuous infusion
Drug: Antithrombin III, Intermittent infusion — Antithrombin-III is administered intermittently
  Other Names: Antithrombin III, human
  Arms: Intermittent infusion

SUMMARY:
This study was designed to demonstrate more effective administration method of AT-III in immediate post-liver transplantation period.

DETAILED DESCRIPTION:
Antithrombin III(AT-III) concentrates have been used to prevent critical thrombosis in the immediate post-liver transplantation period without clear evidence regarding the optimal dose or administration scheme.

The investigators retrospectively analyzed the clinical data from the patients who received liver transplantation and developed pharmacokinetic model of AT-III in the previous research. According to this study, optimal AT-III activity level will be well-maintained with smaller dose with continuous infusion than with intermittent infusion which is widely accepted way of administration currently.

A prospective study was planned to show the more effective manner of AT-III concentrate administration after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled operation
* Living donor liver transplantation
* Adult patients (>=18 years old)

Exclusion Criteria:

* Patients under 18 years old
* Emergency operation
* Deceased donor liver transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients within target range at postoperative 72 hours | 72 hours after liver transplantation
  Proportion of patients whose AT-III activity level is within the target range (80-120%)

SECONDARY OUTCOMES:
Proportion of patients within target range at postoperative 12/24/48/84 hours | 12/24/48/84 hours after liver transplantation
  Proportion of patients whose AT-III activity level is within the target range (80-120%)
Proportion of AT-III level values within target range | 12/24/48/72/84 hours after liver transplantation
  Among the measured AT-III activity levels, proportion of the values within the target range (80-120%)
Time required for AT-III level value to fall within target range | operation day ~ postoperative day 7
  Time required for AT-III level value to fall within target range (80-120%, hours)
Duration for cessation of AT-III concentrate administration | operation day ~ postoperative day 7
  AT-III infusion is stopped for 24 hours when AT-III plasma activity level exceeds 120%, then restarted after the value is confirmed to be less than 120%.
Bleeding requiring intervention | operation day ~ postoperative day 7
  Bleeding requiring intervention
Thrombosis event | operation day ~ postoperative day 7
  Hepatic artery thrombosis, portal vein thrombosis
Postoperative hospital stay | through the hospital day, an average of 14 days
  number of days from operation to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ho Geol Ryu, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea